CLINICAL TRIAL: NCT07199205
Title: Hyperuricemia as a Predictor of Chronic Kidney Disease (CKD) Progression in Prediabetic Patients
Brief Title: Hyperuricemia as Early Indication of CKD Progressing in Prediabetic
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherry Refaat, Resident doctor in Internal medicine department, Assiut University
Other Study IDs: CKD progression in prediabetic
Record Dates: First submitted 2025-09-19; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: CKD Progression
Keywords: CKD; Prediabetes; Hyperuricemia
MeSH Terms: conditions — Prediabetic State; Hyperuricemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: includes individuals at high risk of chronic kidney disease (prediabetic patient s)
- Group 2: individuals diagnosed with early ckd stage A1,A2,A3
- Group 3: serves as the control group and includes participants with normal renal function.

SUMMARY:
Chronic kidney disease (CKD) is a major global health problem, and hyperuricemia has emerged as both a consequence and a potential driver of its progression. Elevated uric acid contributes to renal impairment through oxidative stress, endothelial dysfunction, inflammasome activation, and crystal deposition. Epidemiological studies show that hyperuricemia often precedes CKD and serves as an independent predictor, with prevalence reaching up to 38% among CKD patients.

Prediabetes, another growing health concern, is associated with higher serum uric acid levels and increased risk of developing both diabetes and CKD. Factors such as obesity, fatty liver, and dyslipidemia mediate this link. Clinically, higher uric acid levels are correlated with faster eGFR decline and higher risk of ESRD, with the uric acid/HDL ratio proposed as a novel risk marker.

Although debate persists about whether hyperuricemia directly causes CKD, emerging genetic and epidemiological evidence supports its independent role. Given the rising prevalence of prediabetes and hyperuricemia, identifying hyperuricemia as a modifiable early predictor of CKD progression in prediabetic patients could help improve prevention, risk stratification, and management

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a global health concern, characterized by a gradual loss of kidney function, and is associated with increased morbidity and mortality. Hyperuricemia, defined as elevated serum uric acid levels, has been identified as both a consequence and a potential contributor to CKD progression. Recent studies have shown that hyperuricemia can aggravate renal impairment through mechanisms such as direct nephrotoxicity, activation of the inflammasome, increased oxidative stress, and endothelial dysfunction.

Epidemiological evidence indicates that hyperuricemia often precedes the development of CKD and may serve as an independent predictor of its onset and progression, even after adjusting for traditional risk factors like hypertension, proteinuria, and dyslipidemia. The prevalence of hyperuricemia is notably higher among CKD patients, reaching up to 38% in some populations. Furthermore, hyperuricemia is implicated in the pathogenesis of several metabolic disorders, including hypertension, obesity, and metabolic syndrome, all of which are risk factors for CKD.

Prediabetes, a state of impaired glucose metabolism, is increasingly recognized as a risk factor for both cardiovascular disease and CKD. Studies have found that individuals with prediabetes exhibit higher serum uric acid levels compared to normoglycemic individuals, and that elevated uric acid is associated with increased risk of progression to diabetes and CKD. The relationship between hyperuricemia and prediabetes appears to be mediated by factors such as fatty liver, dyslipidemia, and body mass index, highlighting the complex interplay between metabolic health and kidney function.

Clinical research has demonstrated that higher serum uric acid levels are associated with a more rapid decline in estimated glomerular filtration rate (eGFR) and an increased risk of progression to end-stage renal disease (ESRD). For example, a baseline uric acid level of ≥7.5 mg/dL has been shown to significantly increase the risk of renal function decline in hypertensive and non-diabetic populations. Additionally, the serum uric acid to high-density lipoprotein (HDL) cholesterol ratio has emerged as a novel marker for predicting CKD risk, reflecting the balance between pro-inflammatory and anti-inflammatory processes.

Despite these associations, the causality of hyperuricemia in CKD progression remains a topic of debate, as some clinical trials have yielded conflicting results regarding the benefits of uric acid-lowering therapy in slowing CKD progression. However, recent genetic and epidemiological studies suggest that hyperuricemia represents a significant risk factor for CKD, independent of genetic predisposition and other comorbidities. The mechanisms by which uric acid may induce kidney injury include crystal deposition, oxidative stress, activation of the renin-angiotensin-aldosterone system, and impairment of endothelial function.The burden of CKD in prediabetic individuals is of particular concern, as early identification of modifiable risk factors such as hyperuricemia could facilitate timely interventions to prevent or delay CKD progression. Given the increasing prevalence of both prediabetes and hyperuricemia worldwide, understanding their interplay is crucial for developing effective preventive strategies.

Despite growing evidence linking hyperuricemia to CKD progression, particularly in at-risk populations such as prediabetic patients, the predictive value of elevated serum uric acid for CKD progression in this group remains underexplored. This study aims to clarify whether hyperuricemia can serve as an early and independent predictor of CKD progression in prediabetic patients, thereby informing clinical practice and guiding risk stratification and management in this vulnerable population

ELIGIBILITY:
Inclusion criteria:

* Adults aged 18 years and older.
* Diagnosed with prediabetes, defined according to the American Diabetes - - - - Association (ADA) criteria (fasting plasma glucose 100-125 mg/dL, HbA1c 5.7-6.4%, or 2-hour plasma glucose 140-199 mg/dL after oral glucose tolerance test).
* Baseline estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m² (CKD stages 1-2).
* Willingness to provide informed consent and comply with study procedures.

Exclusion criteria:

* Diagnosis of diabetes mellitus (fasting plasma glucose ≥126 mg/dL, HbA1c ≥6.5%).
* Established CKD stage 3 or higher (eGFR <60 mL/min/1.73 m²).
* History of gout or current use of uric acid-lowering therapy (e.g., allopurinol, febuxostat) or acute gout.
* Use of medications known to significantly affect uric acid levels (e.g., thiazide diuretics, high-dose aspirin).
* Pregnancy or lactation.
* Presence of severe comorbid conditions (e.g., malignancy, active infection, advanced liver disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population divided into three groups:
  The first group includes individuals at high risk of chronic kidney disease (prediabetic patient s) The second group comprises individuals diagnosed with early ckd stage A1,A2,A3 The third group serves as the control group and includes participants with normal renal function
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
CKD progression in prediabetics | 1 year
  Progression of CKD, defined as a sustained reduction in eGFR of ≥25% from baseline or advancement to a higher CKD stage (KDIGO classification) during the follow-up period.

REFERENCES:
- [Background] Johnson MR, Costanzo-Nordin MR, Heroux AL, Kao WG, Mullen GM, Pifarre R, Sullivan HJ. High-risk cardiac operation: a viable alternative to heart transplantation. Ann Thorac Surg. 1993 Apr;55(4):876-82. doi: 10.1016/0003-4975(93)90109-u. PMID 8466342
- [Background] Petro WG, Kendelewicz T, Lindau I I, Spicer WE. Au-GaAs(110) interface: Photoemission studies of the effects of temperature. Phys Rev B Condens Matter. 1986 Nov 15;34(10):7089-7106. doi: 10.1103/physrevb.34.7089. No abstract available. PMID 9939362
- [Background] Bignardi PR, Ido DH, Garcia FAL, Braga LM, Delfino VDA. Does uric acid-lowering treatment slow the progression of chronic kidney disease? A meta-analysis of randomized controlled trials. Nefrologia (Engl Ed). 2023 Mar-Apr;43(2):167-181. doi: 10.1016/j.nefroe.2022.04.005. Epub 2022 Dec 21. PMID 36564223
- [Background] Srivastava A, Kaze AD, McMullan CJ, Isakova T, Waikar SS. Uric Acid and the Risks of Kidney Failure and Death in Individuals With CKD. Am J Kidney Dis. 2018 Mar;71(3):362-370. doi: 10.1053/j.ajkd.2017.08.017. Epub 2017 Nov 11. PMID 29132945
- [Background] Galan I, Goicoechea M, Quiroga B, Macias N, Santos A, Garcia de Vinuesa MS, Verdalles U, Cedeno S, Verde E, Perez de Jose A, Garcia A, Luno J. Hyperuricemia is associated with progression of chronic kidney disease in patients with reduced functioning kidney mass. Nefrologia (Engl Ed). 2018 Jan-Feb;38(1):73-78. doi: 10.1016/j.nefro.2017.04.006. Epub 2017 Aug 30. English, Spanish. PMID 28869042
- [Background] Johnson RJ, Sanchez Lozada LG, Lanaspa MA, Piani F, Borghi C. Uric Acid and Chronic Kidney Disease: Still More to Do. Kidney Int Rep. 2022 Dec 5;8(2):229-239. doi: 10.1016/j.ekir.2022.11.016. eCollection 2023 Feb. PMID 36815099
- [Background] Hung YH, Huang CC, Lin LY, Chen JW. Uric Acid and Impairment of Renal Function in Non-diabetic Hypertensive Patients. Front Med (Lausanne). 2022 Jan 24;8:746886. doi: 10.3389/fmed.2021.746886. eCollection 2021. PMID 35141237
- [Background] Alqahtani SAM, Awan ZA, Alasmary MY, Al Amoudi SM. Association between serum uric acid with diabetes and other biochemical markers. J Family Med Prim Care. 2022 Apr;11(4):1401-1409. doi: 10.4103/jfmpc.jfmpc_1833_21. Epub 2022 Mar 18. PMID 35516683
- [Background] Echouffo-Tcheugui JB, Narayan KM, Weisman D, Golden SH, Jaar BG. Association between prediabetes and risk of chronic kidney disease: a systematic review and meta-analysis. Diabet Med. 2016 Dec;33(12):1615-1624. doi: 10.1111/dme.13113. Epub 2016 Apr 24. PMID 26997583
- [Background] Beaucher WN. How the wheels of "justice" nearly destroyed an innocent doctor. Med Econ. 1993 Nov 22;70(22):170-6. No abstract available. PMID 10130409